CLINICAL TRIAL: NCT03182231
Title: Visualizing Beta Cells in Patients With T2D Before and After Bariatric Surgery
Brief Title: GLP1-imaging Before and After Bariatric Surgery
Status: Unknown | Phase: Phase 1 / Phase 2 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Radboud University Medical Center (Other)
Collaborators: Rijnstate Hospital (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Sequential | Masking: None | Purpose: Basic Science
Other Study IDs: NL51980.091.15
Record Dates: First submitted 2017-05-29; First posted 2017-06-09 (Actual); Last update posted 2022-06-21 (Actual); Status verified 2021-06

CONDITIONS: Diabetes Mellitus, Type 2; Bariatric Surgery Candidate
Keywords: exendin; GLP1; beta cell mass
MeSH Terms: conditions — Diabetes Mellitus, Type 2

STUDY DESIGN:
Intervention Model Description: Patients will receive an 68Ga-NODAGA-exendin-4 PET/CT scan before RYGB and 1 year after RYGB
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- RYGB patients (Experimental): Patients who will receive a RYGB surgery
  Interventions: Radiation: 68Ga-NODAGA-exendin-4 PET/CT

INTERVENTIONS:
Radiation: 68Ga-NODAGA-exendin-4 PET/CT — 68Ga-NODAGA-exendin-4 PET/CT

SUMMARY:
In order to evaluate the difference in beta cell mass in morbidly obese patients with type 2 diabetes mellitus (T2D) before and after Roux-en-Y gastric bypass (RYGB), investigators aim to compare quantitative PET imaging of the pancreas in this patient group before and after surgery. Investigators propose to measure the uptake of 68Ga-NODAGA-exendin-4 in the pancreatic beta cells of these patients. Furthermore, investigators aim to compare uptake of the radiolabeled tracer to beta cell function measured by laboratory parameters. These highly relevant data will provide investigators with more information on the contribution of the beta cells to the mechanisms behind resolution of T2D after bariatric surgery and on the prognostic value of pre-operative beta cell mass determination to T2D resolution. This might be of great interest for the assessment of RYGB as an alternative therapy in patients with T2D and a BMI <35, who currently do not meet the international guidelines for bariatric surgery.

DETAILED DESCRIPTION:
The prevalence of Type 2 Diabetes Mellitus (T2D) in the Netherlands is 600.000-800.000 and each year ~70.000 new patients are diagnosed. This increasing number of patients with T2D is closely correlated with the obesity epidemic.

Obese patients with T2D are also at risk to develop dyslipidemia and hypertension. This clustering of cardiovascular risk factors leads to an increased risk of micro-and macrovascular long-term complications. In fact, patients with T2D have a 2-4 times increased risk for cardiovascular disease. These complications seriously decrease the quality of life and life expectancy of T2D patients. The burden of this disease affects our society as well. Health care costs with respect to diabetes amounted 814 million euro in 2005 in the Netherlands and indirect costs because of absence of work are unknown but thought to be substantial.

Weight loss is perhaps the most important therapeutic intervention in obese patients with T2D. Weight loss intervenes in the underlying pathophysiology and restores insulin sensitivity and sometimes even insulin secretion. In addition, it improves dyslipidemia and hypertension. In contrast, most pharmacological interventions only relieve the symptoms of the complex disease process underlying T2D whilst the disease process itself is not addressed and even progresses in the course of time. Unfortunately, the effect of weight loss interventions such as diet and lifestyle or even drugs (orlistat, sibutramine) is often modest (3-5 kg) and short-lived.

Bariatric surgery and T2D remission Weight reducing surgery, i.e. bariatric surgery, is the only intervention that leads to persistent weight loss and is superior above conventional (non-surgical) treatment. Bariatric surgery can be divided into restrictive (gastric band or sleeve) and malabsorptive (biliopancreatic diversion, BD) procedures or a combination of both (Roux-en-Y gastric bypass, RYGB). Currently, RYGB is the most performed bariatric procedure. The international indications for bariatric surgery are BMI > 40kg/m2 or BMI > 35 kg/m2 with co-morbidities (e.g. T2D).

Besides weight loss, spectacular metabolic improvements after bariatric surgery are seen. In patients with T2D, normalization of fasting plasma glucose and/or HbA1c without medication (referred as "resolution of T2D") was observed in 48% and 83% after gastric banding and RYGB, respectively. Recently, randomized controlled trials showed the superiority of bariatric surgery in glycemic control above conventional medical treatment. Furthermore, the improvement in glycemic control is higher in RYGB compared to purely restrictive bariatric procedures.

The mechanism of diabetes resolution after RYGB is not completely understood and there is evidence that it might not be dependent on weight loss only. Improvements in glycemic control have been found within days after surgery, while significant weight loss has not yet been achieved at this time. There are several hypotheses concerning the weight-independent effects of bariatric surgery on insulin secretion. The most popular are the 'hindgut-hypothesis', which states that expedited delivery of nutrients to the distal intestine enhances the secretion of intestinal peptides like glucagon-like-peptide 1 (GLP1) and peptide YY and the 'foregut hypothesis', which states that the exclusion of the duodenum and proximal jejunum from the transit of nutrients results in changes in secretion of intestinal peptides. However, several other mechanisms, both in- and outside the intestines might play a role.

The beta cell function improves after RYGB in individuals with and without T2D, however it is unclear whether the actual beta cell mass is subject to change after bariatric surgery. Examination of the beta cell mass on autopsy specimens of persons who did not have bariatric surgery, showed a decrease in beta cell mass in persons with T2D in one of the studies a decrease was found in persons with pre-diabetes as well.

Few studies were performed that assessed beta cell mass after bariatric surgery. In Goto-Kakizaki rats duodenal jejunal bypass was found to increase pancreatic concentrations of vesicular monoamine transporter type 2 (VMAT2). VMAT2 was used as a biomarker for beta cells, however later VMAT2 was found to be expressed on pancreatic polypeptide cells (PP cells) as well. Furthermore, an increase in beta cell mass, beta cell number and extra islet beta cells was found after RYGB in a porcine model and GK rat model. Studies in humans showed conflicting results. Long term after gastric bypass, cases of hyperinsulinemic hypoglycemia have been described, which are related to pancreatic islet hyperplasia or nesidioblastosis, while this does not occur after purely restrictive surgery. However, beta cell mass was assessed in six patients after gastric bypass by histological analysis of the pancreas after pancreatectomy and did not find an increase in beta cell mass. These studies were performed on pancreas specimen and not in vivo.

The benefit of RYGB on glycemic control in morbid obese patients (BMI > 35 kg/m2) with T2D is confirmed and the Diabetes Surgery Summit Consensus Conference accepted bariatric surgery as alternative therapy of obesity related T2D. They also consider expanding the indication for bariatric surgery in obese patients with T2D who currently don't meet the international guidelines for bariatric surgery. In this regard it would be helpful to identify preoperatively which T2D patients would benefit from RYGB. Prognostic factors that were described previously are the duration of diabetes, age, preoperatively HbA1c levels and fasting C-peptide. However, the underlying cause of T2D resolution and the prognostic value of these factors are not completely understood. Possibly, T2D resolution depends on the preoperative available beta cell mass and function and increased beta cell failure or reduced beta cell ass might decrease the chance of T2D resolution. Therefore, more information on the effects of bariatric surgery on beta cell function and beta cell mass will be helpful to further understand T2D resolution and the role of the beta cells. Thereby, preoperative beta cell mass might be a prognostic factor of T2D resolution and helpful in identifying obese T2D patients that will benefit from RYGB and expanding the indications for bariatric surgery for those patients. For this purpose reliable, sensitive and specific visualization of living pancreatic beta cells in vivo is important.

GLP-1 receptor imaging by PET For specific non-invasive imaging of beta cells, we have developed a highly beta cell-specific radiolabeled exendin-based GLP-1 analog which, after radiolabeling, can non-invasively be detected in the human body. GLP-1 is an incretin hormone that specifically binds to beta cells and is responsible for post-prandial insulin-secretion. Its specificity for beta cells has been shown and a linear correlation of the beta cell mass and the signal obtained with this tracer has been established.

GLP-1R imaging has been shown to be suitable for imaging of insulin producing pancreatic neuroendocrine tumours (IPPNET). Furthermore, the feasibility of visualization of transplanted beta cells with GLP-1R imaging has been shown by imaging of autologous islets transplanted into muscle.

ELIGIBILITY:
Inclusion Criteria:

* Morbid obese T2D patient who will have RYGB at the Rijnstate in Arnhem
* Female
* Signed informed consent

Mild T2D:

* C-peptide > 1.0 nmol/L
* Only metformin usage as anti-diabetic medication

Progressive T2D:

* C-peptide < 1.0 nmol/L
* Insulin and/or sulfonylurea (SU) usage

Exclusion Criteria:

* Fasting glucose < 6 at time C-peptide was determined
* Liver failure
* BMI > 50 kg/m-2
* Previous treatment with synthetic exendin
* Pregnancy
* Breast feeding
* Kidney failure
* Age < 18 years
* No signed informed consent

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 12 (Estimated)
Dates: Start 2016-10-07 (Actual); Primary Completion 2023-07-01 (Estimated); Study Completion 2023-07-01 (Estimated)

PRIMARY OUTCOMES:
Pancreatic uptake of 68Ga-NODAGA-exendin-4 | 4 years
  Change in tracer uptake before and after RYGB

SECONDARY OUTCOMES:
T2D outcome | after 1 year
  Comparison of tracer uptake with T2D outcome
Beta cell function | 4 years
  Correlation between tracer uptake and beta cell function

CONTACTS AND LOCATIONS:
Locations (2):
- Netherlands (2):
  - Rijnstate hospital, Arnhem
  - Radboudumc, Nijmegen

IPD SHARING:
Plan to Share IPD: No